Identity: AİBÜ-HEM-HHT-01

**Document Date:** September 27, 2022

**Operating protocol** 

Study Title: The Effect of Creative Drama Training for Alcohol-Substance Addicted Male

Patients on Their Attitudes Regarding Violence Against Women: A Randomized Controlled

Study.

**Short title:** Violence Against Women in Patients With Alcohol Substance Addiction Training

There is no NCT number and no discharge.

**Purpose of the Research** 

This study was planned as a randomized controlled trial in order to determine the effect of

creative drama training for alcohol-substance dependent male patients on their attitudes towards

violence against women.

Hypotheses

H0: There was no difference between the attitude scores of the experimental and control groups

on violence.

H0-1: There is no difference between the experimental and control group pretest scores.

H0-2: There is no difference between the final test scores of the experimental and control

groups.

H0-3: There is no difference between the experimental group pretest-posttest scores

H0-4: There is no difference between control group pretest and posttest scores.

## Type of research

This study was designed as a randomized controlled experimental study.

#### Power of research

When there is a difference between two applications, the possibility of revealing this difference is the power of research. In order to make an important inference, this rate must be accepted as at least 80%. In this study, the power of the research was determined as 99%.

# Type 1 error

While there is no difference between the two applications, the difference is found as a result of the research. It is known as the  $\alpha$  or p value. When calculating the sample size, type 1 error is generally accepted as 0.05 or 0.01. The type 1 error amount of this study was accepted as 1%.(74)

# **Impact size**

It is the difference between the value tried to be estimated in the sample of the research and the previously known value of this value in the society and this difference should be determined in advance. As the effect size increases, the number of samples decreases. When the effect size of this study was calculated by referencing the final test scores of the experiment-control group of another study in which this measurement tool was used, the effect size was determined as 1.93.

## Calculation of sample size

As a calculation tool, the G-Power 3.1.9.4 program was used. The effect size of the study was calculated as 1.93, the alpha margin of error: 0.01, the strength as 0.99 and the sample size: 34 for the three groups. Groups; n=17, Considering that there may be a loss of sample, 40 people-experiment: n=20, control: n=20- were included in this study.

## Implementation of Research

It is stated that the research is not mandatory for the participants, that a training on violence against women will be applied and that they can be separated at any stage of the application. The study group consisted of 40 patients diagnosed with alcohol and substance abuse. To prevent interaction, the first application was applied to the control group (n=20). No training was applied to the control group. The pre-test was applied and the final test was applied 9 days later. During this nine-day period, three patients were discharged and the control group was completed with n=17 patients. The second application was applied to the experimental group. Violence against women education was applied to the experimental group through creative drama. The training content is divided into five sessions. SAMBA (Smoking, Alcohol and Substance Abuse Treatment Program) training applied in the process of addiction treatment and psycho-drama studies applied in different subjects are applied every other day considering the hospitalization period of the patients (~21-24 days). Similarly, these trainings were applied

every other day and the final test was applied at the end of the 5th session. At the end of all applications, brochures on "violence against women" were given to the control group and a presentation was made by the researcher. (Ögel K, 2012; Auspicious et al., 2020) "Personal Information Form" and "Violence Against Women Attitude Scale" were applied as pre-tests to the control and experimental group. Participants were told that all questions should be filled in completely.

#### Randomization and Blindness of Research

In this study, the names of the patients hospitalized in the two wards will be sorted and numbered in alphabetical order. After the numbering process, patients will be divided into an experimental and control group using the "https://www.randomizer.org/" site by an independent specialist.

### Ethical dimension of the research

Permission will be obtained from the person to whom the research will be conducted. Written permissions were obtained from the institution where the research will be conducted. Bolu Abant İzzet Baysal University Clinical Research Ethics Committee has received permission numbered 2022-131.

## Analysis of the data

The analysis of the data will be carried out by using SPSS-22 (Statistical Package for Social Sciences) package program. In the evaluation of the data on the descriptive characteristics of the participants, the number, percentage, mean and standard deviation will be used to determine the Attitude scores of the individuals in the experimental and control groups. The Wilcoxon Marked Ranks test will be used to determine whether there is a difference between the participants' scores on the pretest and the post-test "Violence Against Women Attitude Scale". The Mann-Whitney U test will also be used to compare the attitudes of the individuals in the

experimental and control groups as the intergroup pretest-posttest "Violence Against Women Attitude Scale" < 0.05.